CLINICAL TRIAL: NCT02725437
Title: A Phase 1, Placebo-controlled, Randomized, Observer-blinded Study To Evaluate The Safety, Tolerability, And Immunogenicity Of Two 3-dose Regimens Of Clostridium Difficile Vaccine Administered In Healthy Japanese Adults Aged 65 To 85 Years.
Brief Title: Clostridium Difficile Vaccine Safety, Tolerability, and Immunogenicity Study in Japanese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: B5091010
Record Dates: First submitted 2016-01-29; First posted 2016-04-01 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Clostridium Difficile Associated Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Low-dose C. difficile Vaccine (accelerated schedule) (Experimental)
  Interventions: Biological: Clostridium difficile Vaccine
- High-dose C. difficile Vaccine (accelerated schedule) (Experimental)
  Interventions: Biological: Clostridium difficile Vaccine
- Placebo (accelerated schedule) (Placebo Comparator)
  Interventions: Biological: Placebo
- Low-dose C. difficile Vaccine (non-accelerated schedule) (Experimental)
  Interventions: Biological: Clostridium difficile Vaccine
- High-dose C. difficile Vaccine (non-accelerated schedule) (Experimental)
  Interventions: Biological: Clostridium difficile Vaccine
- Placebo (non-accelerated schedule) (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Clostridium difficile Vaccine — 0.5 mL intramuscular injection
  Arms: High-dose C. difficile Vaccine (accelerated schedule); High-dose C. difficile Vaccine (non-accelerated schedule); Low-dose C. difficile Vaccine (accelerated schedule); Low-dose C. difficile Vaccine (non-accelerated schedule)
Biological: Placebo — 0.5 mL intramuscular injection
  Arms: Placebo (accelerated schedule); Placebo (non-accelerated schedule)

SUMMARY:
The first-in-Japanese study B5091010 has been designed to evaluate the safety, tolerability, and immunogenicity of 2 antigen dose levels of C difficile vaccine when administered as one of two 3-dose regimens to healthy Japanese adults aged 65 to 85 years.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female adults
2. Aged 65 to 85 years

Exclusion Criteria:

1. Proven or suspected prior episode of Clostridium difficile associated diarrhea
2. Unstable chronic medical condition
3. Disease requiring significant change in therapy or hospitalization for worsening disease within 8 weeks before receipt of study vaccine
4. Serious chronic medical disorders
5. Bleeding diathesis or condition associated with prolonged bleeding time that may contraindicate intramuscular injection
6. Any contraindication to vaccination or vaccine components, including previous anaphylactic reaction to any vaccine or vaccine-related components
7. Subjects with congenital or acquired immunodeficiency disorders
8. Subjects with rheumatologic disorders or other illnesses requiring chronic treatment with known immunosuppressant medications
9. Active or treated leukemia or lymphoma or bone marrow disorder
10. Residence in a nursing home or other long-term care facility, or requirement for semiskilled nursing care or assisted living
11. Abnormality in screening hematology and/or blood chemistry laboratory values

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Proportions of subjects reporting local reactions (pain, erythema, and induration) and their severity, as self-reported on e-diaries | Up to 14 days after each vaccination
Proportions of subjects reporting systemic events (fever, vomiting, diarrhea, headache, fatigue, new or worsening muscle pain, and new or worsening joint pain) and their severity, as self-reported on e-diaries | Up to 14 days after each vaccination
Proportions of subjects reporting AEs (categorized according to the Medical Dictionary for Regulatory Activities [MedDRA]) | From the first vaccination up to 28 days after the last vaccination
Proportions of subjects reporting SAEs (categorized according to the Medical Dictionary for Regulatory Activities [MedDRA]) | From the first vaccination until 6 months after the last vaccination
Proportions of subjects with abnormal hematology and blood chemistry laboratory assessments | 7 days or 14 days after each vaccination

SECONDARY OUTCOMES:
Toxin A- and toxin B-specific neutralizing antibody levels, expressed as geometric mean concentrations | Up to 6 months after dose 3
Geometric mean fold rises in toxin A- and toxin B-specific neutralizing antibody levels | Up to 6 months after dose 3
Proportions of subjects in each vaccine group with toxin A-specific neutralizing antibody level ≥ the specified threshold for toxin A | Up to 6 months after dose 3
Proportions of subjects in each vaccine group with toxin B-specific neutralizing antibody level ≥ the specified threshold for toxin B | Up to 6 months after dose 3
Proportions of subjects in each vaccine group with both toxin A- and toxin B-specific neutralizing antibody levels ≥ the specified threshold for toxin A and the specified threshold for toxin B, respectively | Up to 6 months after dose 3
Proportions of subjects in each vaccine group with fold rises in toxin A-specific neutralizing antibody levels | Up to 6 months after dose 3
Proportions of subjects in each vaccine group with fold rises in toxin B-specific neutralizing antibody levels | Up to 6 months after dose 3
Proportions of subjects in each vaccine group with fold rises in both toxin A- and toxin B-specific neutralizing antibody levels | Up to 6 months after dose 3

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Japan (2):
  - SOUSEIKAI Sumida Hospital (formerly Medical Co. LTA Sumida Hospital), Sumida-ku, Tokyo
  - SOUSEIKAI PS Clinic (formerly Medical Co. LTA PS Clinic), Fukuoka

REFERENCES:
- [Derived] Inoue M, Yonemura T, de Solom R, Yamaji M, Aizawa M, Knirsch C, Pride MW, Jansen KU, Gruber W, Webber C. A phase 1 randomized study assessing safety and immunogenicity of two 3-dose regimens of a Clostridium difficile vaccine in healthy older Japanese adults. Vaccine. 2019 May 1;37(19):2600-2607. doi: 10.1016/j.vaccine.2019.03.014. Epub 2019 Apr 5. PMID 30962095
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5091010&StudyName=A%20Phase%201%2C%20Placebo-controlled%2C%20Randomized%2C%20Observer-blinded%20Study%20To%20Evaluate%20The%20Safety%2C%20Tolerability%2C%20And%20Immunogenicity%20Of%20Two%203-dose%20Regimens%20Of%20Clostridium%20Difficile%20Vaccine%20Administered%20In%20Healthy%20Japanese%20Adults%20Aged%2065%20To%2085%20Years.
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5091010&StudyName=A+Phase+1%2C+Placebo-controlled%2C+Randomized%2C+Observer-blinded+Study+To+Evaluate+The+Safety%2C+Tolerability%2C+And+Immunogenicity+Of+Two+3-dose+Regimens+Of+Clostridium+Difficile+Vaccine+Administered+In+Healthy+Japanese+Adults+Aged+65+To+85+Years.